CLINICAL TRIAL: NCT04270682
Title: A Phase 3 Study to Evaluate the Effects of Chenodeoxycholic Acid in Adult and Pediatric Patients With Cerebrotendinous Xanthomatosis
Brief Title: Study to Evaluate Patients With Cerebrotendinous Xanthomatosis (RESTORE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cheno-CTX-301
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: CTX
Keywords: Cerebrotendinous xanthomatosis; CTX; Cholestanol; Leukodystrophy; CYP27A1
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous

STUDY DESIGN:
Intervention Model Description: Two-cohort study. One cohort is for adult patients with a double-blind placebo withdrawal (with CDCA rescue) crossover. Second cohort will dose titrate pediatric patients into a stable, open-label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult Cohort (Experimental): Patients in the adult cohort will participate in a randomized, double-blind, placebo-controlled, 2 period × 2-treatment crossover study with rescue medication and open-label run-in to assess the efficacy and safety of CDCA.
  Interventions: Drug: Blinded CDCA 250 mg TID; Drug: Placebo; Drug: Open-Label CDCA 250 mg TID; Drug: Rescue Medication CDCA 250 mg TID
- Pediatric Cohort (Experimental): Pediatric cohort patients (≥1 month and <16 years) will participate in a 24-week, open-label cohort with an 8-week titration period and a 16-week treatment period at the tolerated dose.
  Interventions: Drug: CDCA Weight-Based Dose TID

INTERVENTIONS:
Drug: Blinded CDCA 250 mg TID — Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Arms: Adult Cohort
Drug: Placebo — Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Arms: Adult Cohort
Drug: Open-Label CDCA 250 mg TID — Adult cohort patients will receive open-label 250 mg CDCA TID during the run-in and washout periods of the study or as rescue medication during the double-blind periods, if needed, based on clinical symptoms.
  Arms: Adult Cohort
Drug: Rescue Medication CDCA 250 mg TID — CDCA 250 mg TID will be provided as rescue medication during the double-blind periods, if needed, based on laboratory results.
  Arms: Adult Cohort
Drug: CDCA Weight-Based Dose TID — Patients in the pediatric cohort will complete a weight-based dose titration to a tolerated dose and will maintain that tolerated dose for the remainder of the study. Pediatric cohort dosing of CDCA will not exceed an equivalent dose of 750 mg/day.
  Arms: Pediatric Cohort

SUMMARY:
The study is made up of two cohorts: a randomized double-blind crossover (placebo withdrawal with rescue) study among patients ≥ 16 years of age (adult cohort) and an open-label dose titration study among pediatric patients ≥1 month and <16 years of age (pediatric cohort)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 1 month or older at screening.
2. Clinical diagnosis of CTX with biochemical confirmation.
3. Women of childbearing potential must agree to the use of one highly reliable method of contraception during the study, plus one additional barrier method during sexual activity.
4. Males must be surgically sterile, or males and their sexual partners must together agree to use medically accepted methods of contraception that are considered highly reliable during the course of the study.

Exclusion Criteria:

1. Genetic testing does not confirm CTX.
2. Malabsorption disorder or confounding inflammatory gastrointestinal condition (for example, irritable bowel syndrome).
3. Documented history of heart failure.
4. Treated with medications which impact bile acid absorption such as bile acid sequestering agents (eg, cholestyramine, colestipol, aluminum-based antacids.
5. Treated with cholic acid medication.
6. Female patient who is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
7. Positive at screening for the human immunodeficiency virus (HIV) or markers indicating acute or chronic hepatitis B infection or hepatitis C infection.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Travere Investigational Site, Aurora, Colorado
  - Travere Investigational Site, Orlando, Florida
  - Travere Investigational Site, Iowa City, Iowa
  - Travere Investigational Site, New Orleans, Louisiana
  - Travere Investigational Site, Great Neck, New York
  - Travere Investigational Site, Columbus, Ohio
  - Travere Investigational Site, Austin, Texas
  - Travere Investigational Site, Seattle, Washington
- Brazil (3):
  - Travere Investigational Site, Fortaleza, Ceará
  - Travere Investigational Site, Porto Alegre, Rio Grande do Sul
  - Travere Investigational Site, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence AB: Patients in the adult cohort participated in a randomized, double-blind, placebo-controlled, 2 period × 2-treatment crossover study with rescue medication and open-label run-in to assess the efficacy and safety of CDCA.
  Patients randomized to sequence AB received blinded 250 mg CDCA TID for DB1 and Placebo TID for DB2.
  Open-Label CDCA 250 mg TID: Adult cohort patients received open-label 250 mg CDCA TID during the run-in and washout periods of the study or as rescue medication during the double-blind periods, if needed, based on clinical symptoms.
  Rescue Medication CDCA 250 mg TID: CDCA 250 mg TID was provided as rescue medication during the double-blind periods, if needed, based on laboratory results.
- Sequence BA: Patients in the adult cohort participated in a randomized, double-blind, placebo-controlled, 2 period × 2-treatment crossover study with rescue medication and open-label run-in to assess the efficacy and safety of CDCA.
  Patients randomized to sequence BA received blinded Placebo TID for DB1 and 250 mg CDCA TID for DB2.
  Open-Label CDCA 250 mg TID: Adult cohort patients received open-label 250 mg CDCA TID during the run-in and washout periods of the study or as rescue medication during the double-blind periods, if needed, based on clinical symptoms.
  Rescue Medication CDCA 250 mg TID: CDCA 250 mg TID was provided as rescue medication during the double-blind periods, if needed, based on laboratory results.
- Pediatric Cohort: Pediatric cohort patients (≥1 month and <16 years) participated in a 24-week, open-label cohort with an 8-week titration period and a 16-week treatment period at the tolerated dose.
  CDCA Weight-Based Dose TID: Patients in the pediatric cohort completed a weight-based dose titration to a tolerated dose and maintained that tolerated dose for the remainder of the study. Pediatric cohort dosing of CDCA was not to exceed an equivalent dose of 750 mg/day.
Period: Overall Study
Arm/Group | Sequence AB | Sequence BA | Pediatric Cohort
Started | 6 | 7 | 5
Completed | 6 | 7 | 4
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adult Cohort: Start of Run-In Period [Day-56/R1W1, First Day] Pediatric Cohort: Start of Treatment (Day 1)
Groups:
- Sequence AB: Patients in the adult cohort will participate in a randomized, double-blind, placebo-controlled, 2 period × 2-treatment crossover study with rescue medication and open-label run-in to assess the efficacy and safety of CDCA.
  Patients randomized to sequence AB will receive blinded CDCA TID for 4 weeks or until open-label rescue medication criteria are triggered
  Blinded CDCA 250 mg TID: Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Placebo: Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Open-Label CDCA 250 mg TID: Adult cohort patients will receive open-label 250 mg CDCA TID during the run-in and washout periods of the study or as rescue medication during the double-blind periods, if needed, based on clinical symptoms.
- Sequence BA: Patients in the adult cohort will participate in a randomized, double-blind, placebo-controlled, 2 period × 2-treatment crossover study with rescue medication and open-label run-in to assess the efficacy and safety of CDCA.
  Patients randomized to sequence BA will receive placebo TID for 4 weeks or until either the blinded and/or open-label rescue medication criteria are triggered.
  Blinded CDCA 250 mg TID: Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Placebo: Adult cohort patients will receive blinded 250 mg CDCA TID or placebo during the double-blind periods based upon their treatment assignment.
  Open-Label CDCA 250 mg TID: Adult cohort patients will receive open-label 250 mg CDCA TID during the run-in and washout periods of the study or as rescue medication during the double-blind periods, if needed, based on clinical symptoms.
  Rescue Medication CDCA 250 mg TID: CDCA 250 mg TID will be provided as rescue medication during the double-blind periods, if needed, based on laboratory results.
- Total: Total of all reporting groups
Arm/Group | Sequence AB | Sequence BA | Pediatric Cohort | Total
Number analyzed (Participants) | 6 | 7 | 5 | 18
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Thirteen of 14 enrolled participants (92.9%) were randomized and completed the study. One participant was enrolled, but was not randomized, and withdrew from the study.
  years
    Number Analyzed | 43 (7.4) | 38.6 (11.73) | 8.2 (3.96) | 29.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Thirteen of 14 enrolled participants (92.9%) were randomized and completed the study. One participant was enrolled, but was not randomized, and withdrew from the study.
  Participants
    Female | 1 | 4 | 5 | 10
    Male | 5 | 3 | 0 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Thirteen of 14 enrolled participants (92.9%) were randomized and completed the study. One participant was enrolled, but was not randomized, and withdrew from the study.
  Participants
    Asian | 1 | 1 | 0 | 2
    White | 5 | 3 | 5 | 13
    Other | 0 | 2 | 0 | 2
    Multiple | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Population: Thirteen of 14 enrolled participants (92.9%) were randomized and completed the study. One participant was enrolled, but was not randomized, and withdrew from the study.
  participants
    United States | 3 | 4 | 3 | 10
    Brazil | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urine 23S-Pentol During the Two Double-Blind Periods
Description: Primary Analysis of Change from Baseline in Urine 23S-Pentol (Natural Log-Transformed) during the Two Double-blind Periods- Paired T-test
Time Frame: Two double-blind periods: Week 0 to Week 4, Week 12 to Week 16
Population: All adult cohort participants who were randomized and took at least one dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: natural log of ng/mL
Groups:
- CDCA TID: Active: Contains 250 mg of Chenodiol (the non-proprietary name for CDCA). Open-label and blinded CDCA are the same drug product.
- Placebo TID: Control: Placebo study medication is provided in the same form as blinded CDCA, as white film-coated 250-mg tablets with no CDCA.
Arm/Group | CDCA TID | Placebo TID
Number analyzed (Participants) | 13 | 13
natural log of ng/mL
  Pooled Double Blind Baseline | 7.18 (0.797) | 6.96 (1.076)
  Pooled last non missing postbaseline Double Blind record | 7.45 (0.675) | 10.34 (0.788)
  Pooled change from baseline to last non missing postbaseline Double Blind record | 0.20 (0.732) | 3.38 (1.111)
Statistical Analysis 1: Comparison: CDCA TID vs Placebo TID; Test type: Equivalence — The null (H0) hypothesis and the alternative (Ha) hypothesis to be tested for the primary efficacy endpoint are that H0: Δ = 0 versus Ha: Δ ≠ 0 where Δ is the true paired treatment difference between CDCA and placebo for the change from baseline in loge-transformed urine 23S-pentol in the adult cohort; p < 0.0001, paired t-test; Mean Difference (Final Values) = -3.06, 95% CI 2-sided [-3.794 to -2.331], Standard Error of Mean 0.332

2. Secondary Outcome: Change From Baseline Plasma Cholestanol During the Two Double-Blind Periods
Description: Primary Analysis of Change from Baseline Plasma Cholestanol (Natural Log-transformed) at the End of the Two Double-Blind Periods- Paired T-test
Time Frame: Two double-blind periods: Week 0 to Week 4, Week 12 to Week 16
Population: All adult cohort participants who were randomized and took at least one dose of randomized study medication, and who had been on CDCA for at least 2 months prior to the open-label run-in period.
Measure: Mean (Standard Deviation); unit: natural log of μg/mL
Arm/Group | CDCA TID | Placebo TID
Number analyzed (Participants) | 7 | 7
natural log of μg/mL
  Pooled Double Blind baseline | 1.13 (0.791) | 1.14 (0.534)
  Pooled last non missing post baseline Double Blind record | 1.10 (0.728) | 1.88 (0)
  Pooled change from baseline to last non missing post baseline Double Blind record | -0.12 (0.542) | 0.75 (0.865)
Statistical Analysis 1: Comparison: CDCA TID vs Placebo TID; Test type: Equivalence — The null (H0) hypothesis and the alternative (Ha) hypothesis to be tested for the primary efficacy endpoint are that H0: Δ = 0 versus Ha: Δ ≠ 0 where Δ is the true paired treatment difference between CDCA and placebo for the change from baseline in loge-transformed plasma cholestanol in the adult cohort; p = 0.0083, paired t-test; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.640 to -0.399], Standard Error of Mean 0.241

3. Secondary Outcome: Change From Baseline Plasma 7αC4 During the Two Double-Blind Periods
Description: Primary Analysis of Change from Baseline Plasma 7αC4 (Natural Log-Transformed) During the Two Double-Blind Periods
Time Frame: Two double-blind periods: Week 0 to Week 4, Week 12 to Week 16
Population: All adult cohort participants who were randomized and took at least one dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: natural log of ng/mL
Arm/Group | CDCA TID | Placebo TID
Number analyzed (Participants) | 13 | 13
natural log of ng/mL
  Pooled Double Blind baseline | 4.02 (0.519) | 4.00 (0.526)
  Pooled last non missing postbaseline Double Blind record | 3.97 (0.572) | 7.60 (0.511)
  Pooled change from baseline to last non missing postbaseline Double Blind record | -0.08 (0.717) | 3.60 (0.742)
Statistical Analysis 1: Comparison: CDCA TID vs Placebo TID; Test type: Equivalence — The null (H0) hypothesis and the alternative (Ha) hypothesis to be tested for the primary efficacy endpoint are that H0: Δ = 0 versus Ha: Δ ≠ 0 where Δ is the true paired treatment difference between CDCA and placebo for the change from baseline in loge-transformed Plasma 7αC4 in the adult cohort; p < 0.0001, paired t-test; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-4.193 to -3.207], Standard Error of Mean 0.224

4. Secondary Outcome: Proportion of Participants Who Received Rescue Treatment During Two Double-Blind Periods
Description: Proportion of Participants Who Received Rescue Treatment during Two Double-Blind Periods - Prescott's Method
Time Frame: Two double-blind periods: Week 0 to Week 4, Week 12 to Week 16
Population: All adult cohort participants who were randomized and took at least one dose of randomized study medication.
Measure: Number; unit: participants
Arm/Group | CDCA TID | Placebo TID
Number analyzed (Participants) | 13 | 13
participants
  Double Blind Period 1 Proportion of participants who required rescue medication, %: number analyzed (Participants) | 6 | 7
  Double Blind Period 1 Proportion of participants who required rescue medication, % | 0 | 2
  Double Blind Period 2 Proportion of participants who required rescue medication, %: number analyzed (Participants) | 7 | 6
  Double Blind Period 2 Proportion of participants who required rescue medication, % | 1 | 6
  Pooled Proportion of participants who required rescue medication, % | 1 | 8
Statistical Analysis 1: Comparison: CDCA TID; Test type: Equivalence — Exact 2 sided p-value for observing contingency tables of rescue data with equal or more extreme values is calculated using Prescott's method. Rejection of the null hypothesis for no association suggests there is a difference between two treatments; p = 0.0006, Prescott's; proportion = 0.077, 95% CI 2-sided [0.00 to 0.36]
Statistical Analysis 2: Comparison: Placebo TID; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.0006, Prescott's; proportion = 0.62, 95% CI 2-sided [0.32 to 0.86]

ADVERSE EVENTS:
Time Frame: AEs (including SAEs) were captured from the time informed consent was signed to the patient's final visit. In addition, AEs (including SAEs) were to be collected for all patients via a follow-up phone call 30 (±7) days after the last dose of study medication to assess patient safety. Adult Cohort: 24 weeks duration Pediatric Cohort: 16 week duration
Description: * Symptoms described by the patient
  * Clinically significant changes in the patient's physical examination or other signs observed by the Investigator or medical staff
  * Test abnormalities (laboratory tests, ECG, X-rays, etc.) that reflect a change from baseline and/or that may result in changes in administration of study medication or in an alteration in medical care (diagnostic or therapeutic)
  * Conditions present at baseline that have either worsened or recurred following resolution
Groups:
- CDCA: Patients in the adult cohort ; blinded CDCA 250 mg TID in DB1 or DB2
  Treatment-Emergent Adverse Events (TEAEs) were defined as those that start from Open-label Period 1 throughout the study, or existing AEs that worsen during or after Open-label Period 1.
- Placebo: Patients in the adult cohort ; Placebo 250 mg TID in DB1 or DB2
  Treatment-Emergent Adverse Events (TEAEs) were defined as those that start from Open-label Period 1 throughout the study, or existing AEs that worsen during or after Open-label Period 1.
Arm/Group | CDCA | Placebo | Pediatric Cohort
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13 | 0/5
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDCA (N=13) | Placebo (N=13) | Pediatric Cohort (N=5)
Gait Disturbance (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CDCA (N=13) | Placebo (N=13) | Pediatric Cohort (N=5)
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis Viral (Gastrointestinal disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0
Gait Disturbance (General disorders) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aminotransferase Increased (Investigations) | 0 | 0 | 1
Bilirubin Increase (Investigations) | 0 | 1 | 1
Athralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0
Cerebral disorder (Nervous system disorders) | 1 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizzyness (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Blood bilirubin increased (Infections and infestations) | 0 | 1 | 0
Electroencephalogram abnormal (Investigations) | 1 | 0 | 0
Tandem gait test abnormal (Investigations) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0
Lip Infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04270682/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT04270682/SAP_001.pdf